CLINICAL TRIAL: NCT04012619
Title: Safety and Efficacy of Anlotinib Hydrochloride Combined With Pemetrexed Plus Cisplatin/Carboplatin (AP) as First Line Treatment for Stage IIIB/IIIC/IV Non-squamous Non-small-cell Lung Cancer
Brief Title: Anlotinib Hydrochloride Combined With AP in Stage IIIB/IIIC/IV Non-squamous Non-small-cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan University (Other)
Collaborators: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Principal Investigator, You Lu, Chair of Department of Thoracic Cancer, Sichuan University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ALTER-L003
Record Dates: First submitted 2019-07-05; First posted 2019-07-09 (Actual); Results first posted 2023-08-03 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Non-squamous Non-small-cell Lung Cancer; Anlotinib
MeSH Terms: interventions — Pemetrexed

STUDY DESIGN:
Intervention Model Description: The initial dose of anlotinib was set as 12 mg/day with a 2-week on/1-week of schedule. The dose was reduced to 10 mg/day and 8 mg/day in sequence depending on observed DLTs in cycle 1.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Anlotinib Hydrochloride Combined With AP (Experimental): Patients receive pemetrexed (500mg/m2) with cisplatin (75mg/m2)/carboplatin (area under the curve 5) once every 3 weeks, and anlotinib (dose escalation) once daily on days 1-14 of a 21-day cycle. Anlotinib with AP will be administrated up to 4 cycles followed by maintenance treatment with anlotinib once daily (12mg/d) on days 1-14 of a 21-day cycle until disease progression or treatment intolerance.
  Interventions: Drug: Anlotinib Hydrochloride

INTERVENTIONS:
Drug: Anlotinib Hydrochloride — Patients receive pemetrexed with cisplatin/carboplatin once every 3 weeks, and anlotinib (dose escalation) once daily on days 1-14.
  Other Names: Pemetrexed,cisplatin/carboplatin

SUMMARY:
Anlotinib is a novel oral multitarget tyrosine kinase inhibitor and primary targeted to VEGFR, FGFR, PDGFR and c-Kit. The ALTER-0303 trial showed that patients with advanced non-small cell lung cancer (NSCLC) who received anlotinib as third-line or further therapy had more survival benefit. Pemetrexed plus platinum-based chemotherapy (AP) was long considered as the first line treatment in non-squamous NSCLC patients with negative driver mutation. In this dose exploration study, the primary objective is to establish the safety profile of anlotinib combined with AP in non-squamous NSCLC patients by identifying dose limiting toxicity (DLT), maximum tolerance dose (MTD), the recommended phase II dose, and schedule. Secondary objective includes the assessment of preliminary antitumor effect.

DETAILED DESCRIPTION:
Anlotinib, a new small molecule inhibitor of multiple receptor tyrosine kinases targeting the vascular endothelial growth factor receptor (VEGFR), fibroblast growth factor receptor (FGFR), platelet-derived growth factor receptor (PDGFR) and c-Kit,8,9 has been approved as a third-line treatment for refractory advanced NSCLC by the China Food and Drug Administration (CFDA) on May 9, 2018.10 Previous study in phase II (ALTER0302) trial has shown a better progression-free survival (PFS) in advanced NSCLC patients treated with anlotinib compared those with the placebo (4.8 vs 1.2 months, P<0.0001).11 In phase III (ALTER0303) trial, both the overall survival (OS) and PFS of advanced NSCLC patients were observed to be significantly longer in the anlotinib group (median, 9.6 and 5.4 months) than the placebo group (median, 6.3 and 1.4 months).12 Moreover, anlotinib also displayed manageable toxicity, long circulation, and broad-spectrum antitumor potential.13,14 For the lack of recommended drugs with exactly therapeutic effect in the third-line treatment of SCC patients, it is worth to further analyze the efficacy and specifically clinical observation indicator of anlotinib in this subtype of NSCLC patients. In this dose exploration study, the primary objective is to establish the safety profile of anlotinib combined with AP in treatment-naive non-squamous NSCLC patients by identifying dose limiting toxicity (DLT), maximum tolerance dose (MTD), the recommended phase II dose, and schedule. Secondary objective includes the assessment of preliminary antitumor effect.

ELIGIBILITY:
Inclusion Criteria:

* 18 Years to 75 Years patients voluntarily participate in this study, signed and dated informed consent with good compliance and follow-up;
* Diagnosed as locally advanced and / or metastatic non-squamous non-small cell lung adenocarcinoma (NSCLC) by cytology or histology; Provide detectable specimens (tissue or blood) for genotyping before enrollment, and the patients should be with negative EGFR, ALK and ROS1 gene test results, and without prior systemic therapy;
* At least one target lesion that has not received radiotherapy, and has accurate measurement by magnetic resonance imaging (MRI) or computed tomography (CT) (conventional CT≥20 mm or spiral CT≥10 mm) in at least 1 direction;
* Life expectancy is at least 3 months;
* ECOG PS Scoring: 0~1 point;
* The main organs function are normally, the following criteria are met:

  * Blood routine examination criteria (no blood transfusion and blood products within 14 days, no correction by G-CSF and other hematopoietic stimuli):

    i) hemoglobin (HB) ≥90g/L ii) neutrophil absolute (ANC) ≥1.5×109/L iii) platelet (PLT) ≥80×109/L
  * Biochemical tests meet the following criteria i) total bilirubin (TBIL) ≤1.5 times of upper limit of normal (ULN); ii) alanine aminotransferase (ALT) and aspartate aminotransferase (AST)≤2.5 ULN, if liver metastasis occurred, ALT and AST ≤5 ULN; iii) serum creatinine (Cr) ≤1.25 ULN or creatinine clearance (CCr)≥45mL/min (Cockcroft-Gault formula).
* Female patients of childbearing age agree that contraceptive measures must be used within the study period and within 8 weeks after the end of the study drug treatment. The serum or urine test indicates unpregnancy within 7 days prior to the study. Male patients agree to have contraceptive use during the study period and within 8 weeks after the end of the study period or have had surgical sterilization.

Exclusion Criteria:

* Patients with small cell lung cancer (including small cell carcinoma and non-small cell carcinoma mixed lung cancer) and lung adenosquamous carcinoma mixed with squamous carcinoma;
* Active brain metastases, cancerous meningitis, spinal cord compression, or imaging CT or MRI screening for brain or pia mater disease (a patient with brain metastases who have completed treatment and stable symptoms in 21 days before enrollment may be enrolled, but should be confirmed by brain MRI, CT or venography evaluation as no cerebral hemorrhage symptoms);
* Imaging (CT or MRI) shows that the distance between tumor lesion and the large blood vessel is ≤ 5 mm, or there is a central tumor that invades the local large blood vessel and the distance between tumor and bronchial tree is ≤ 2 cm; or there is a significant pulmonary cavity or necrotizing tumor;
* Uncontrollable hypertension (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg after optimal medical treatment);
* Suffering from severe cardiovascular disease: myocardial ischemia or myocardial infarction above grade II, poorly controlled arrhythmias (including men with QTc interval ≥ 450 ms, women ≥ 470 ms); according to NYHA criteria, grades III to IV Insufficient function, or cardiac color Doppler ultrasound examination indicates left ventricular ejection fraction (LVEF) <50%;
* Abnormal blood coagulation (INR > 1.5 or prothrombin time (PT) > ULN + 4 seconds or APTT > 1.5 ULN), with bleeding tendency or undergoing thrombolytic or anticoagulant therapy;
* Urine routine test protein ≥++, and confirmed 24 hours urine protein> 1.0 g;
* There is currently a peripheral neuropathy of ≥CTCAE 2 degrees, except for trauma;
* Respiratory syndrome (≥CTC AE grade 2 dyspnea), serous effusion (including pleural effusion, ascites, pericardial effusion) requiring surgical treatment;
* Long-term unhealed wounds or fractures;
* Serious infection (≥CTC AE Level 2 infection) requiring systemic antibiotics; decompensated diabetes or other ailments treated with high doses of glucocorticoids;
* Active or chronic hepatitis C or/and hepatitis B infection;
* Factors that have a significant impact on oral drug absorption, such as inability to swallow, chronic diarrhea, and intestinal obstruction;
* Patients have undergone major surgery within 4 weeks before enrollment or have severe trauma, fracture and ulcer;
* Severe weight loss (greater than 10%) within 6 weeks prior to enrollment;
* Clinically significant hemoptysis (daily hemoptysis greater than 50ml) within 3 months prior to enrollment; or significant clinically significant bleeding symptoms or defined bleeding tendency, such as gastrointestinal bleeding, hemorrhagic gastric ulcer, baseline fecal occult blood ++ and above, or suffering from vasculitis;
* Events of venous/ arterious thrombosis occurring within the first 12 months prior to enrollment, such as cerebrovascular accidents (including transient ischemic attacks, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism;
* Patients have contraindication to platinum drugs (cisplatin/carboplatin) and cytotoxic drug (Pemetrexed);
* Patients have anaphylactic reaction due to anlotinib Hydrochloride or the excipient in investigational drug.
* Patients have anaphylactic reaction due to contrast agent;
* Planned for systemic anti-tumor therapy during the study period or within 4 weeks prior to enrollment, including cytotoxic therapy, signal transduction inhibitors, immunotherapy (or use mitomycin C within 6 weeks prior to receiving investigational drug). Radiation-rehabilitation radiotherapy (EF-RT) was performed within 4 weeks before enrollment or limited-field radiotherapy was performed for planned tumor lesions within 2 weeks before enrollment.
* Patients were diagnosed with disease which will severely endanger the security of patients or influence the completion of this research, or patients with other situations are not suitable for the study according to the researchers.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2019-11-05 (Actual); Study Completion 2020-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: You Lu, MD, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A standard 3+3 dose reduction design: the initial dose of anlotinib was set as 12 mg/day with a 2-week on/1-week of schedule; the dose was reduced to 10 mg/day and 8 mg/day in sequence depending on observed DLTs in cycle 1. Pemetrexed (500 mg/m2) and either cisplatin (75 mg/m2) or carboplatin (AUC=5) were intravenously given on Day 1 of each cycle.
Groups:
- Anlotinib Hydrochloride (12mg) Combined With AP: Patients receive pemetrexed (500mg/m2) with cisplatin (75mg/m2)/carboplatin (area under the curve 5) once every 3 weeks, and anlotinib (12mg) once daily on days 1-14 of a 21-day cycle. Anlotinib with AP will be administrated up to 4 cycles followed by maintenance treatment with anlotinib once daily (12mg/d) on days 1-14 of a 21-day cycle until disease progression or treatment intolerance.
- Anlotinib Hydrochloride (10mg) Combined With AP: Patients receive pemetrexed (500mg/m2) with cisplatin (75mg/m2)/carboplatin (area under the curve 5) once every 3 weeks, and anlotinib (10mg) once daily on days 1-14 of a 21-day cycle. Anlotinib with AP will be administrated up to 4 cycles followed by maintenance treatment with anlotinib once daily (10mg/d) on days 1-14 of a 21-day cycle until disease progression or treatment intolerance.
Period: Overall Study
Arm/Group | Anlotinib Hydrochloride (12mg) Combined With AP | Anlotinib Hydrochloride (10mg) Combined With AP
Started | 4 | 4
Completed | 4 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Anlotinib Hydrochloride (12mg) Combined With AP; Anlotinib Hydrochloride (10mg) Combined With AP: This dose-exploration study was a standard 3+3 dose reduction design, and eligible patients received an anlotinib chemotherapy regimen after a 21-day cycle for 4 cycles. The initial dose of anlotinib was set as 12 mg/day with a 2-week on/1-week of schedule. The dose was reduced to 10 mg/day and 8 mg/day in sequence depending on observed DLTs in cycle 1. If there were no DLTs, the dose of anlotinib in the combined chemotherapy regimen was determined to be 12 mg/day. If a DLT occurred in≥2 of 3 enrolled subjects, the initial dose was reduced to 10 mg/day. If DLT occurred in 1 of 3 subjects, the dose level was followed up, and 3 additional subjects were enrolled. If 1 DLT occurred in the last 3 subjects, the dose was reduced to 10 mg/day. Pemetrexed (500 mg/m2) and either cisplatin (75 mg/m2) or carboplatin (AUC=5) were intravenously given on Day 1 of each cycle. Patients who had disease control after the combination regimen continued to receive anlotinib maintenance until disease progression was observed.
- Total: Total of all reporting groups
Arm/Group | Anlotinib Hydrochloride (12mg) Combined With AP | Anlotinib Hydrochloride (10mg) Combined With AP | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 2 | 6
  >=65 years | 0 | 2 | 2
Age, Continuous [Median (Full Range); unit: years] | 61 [39 to 62] | 66 [62 to 69] | 62 [39 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 2 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 4 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Smoking history [Count of Participants; unit: Participants]
  Ever | 2 | 2 | 4
  Never | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: the Maximum Tolerated Dose (MTD)
Description: The primary endpoint was the MTD of anlotinib, at which less than 33% of patients experienced a DLT in the frst treatment cycle. A DLT involving hematological toxicity was defned as grade 4 and above, non-hematological toxicity as grade 3 and above, and liver and kidney function injury as grade 2 and above.
Time Frame: 1 month
Measure: Number; unit: mg
Arm/Group | Anlotinib Hydrochloride Combined With AP
Number analyzed (Participants) | 8
mg | 10

ADVERSE EVENTS:
Time Frame: 12 months
Description: Adverse events (AEs) were monitored during the study and summarized according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.0.
Arm/Group | Anlotinib Hydrochloride (12mg) Combined With AP | Anlotinib Hydrochloride (10mg) Combined With AP
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 2/4 | 0/4
Other Adverse Events (participants affected / at risk) | 4/4 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Anlotinib Hydrochloride (12mg) Combined With AP (N=4) | Anlotinib Hydrochloride (10mg) Combined With AP (N=4)
appetite loss (Metabolism and nutrition disorders) | 1 | 0
hand-foot syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Anlotinib Hydrochloride (12mg) Combined With AP (N=4) | Anlotinib Hydrochloride (10mg) Combined With AP (N=4)
Hand-foot syndrome (Musculoskeletal and connective tissue disorders) | 2 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 0
Proteinuria (Gastrointestinal disorders) | 1 | 1
Hypertension (Cardiac disorders) | 3 | 1
Vomiting (Metabolism and nutrition disorders) | 2 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 3
Anemia (Blood and lymphatic system disorders) | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-01): https://cdn.clinicaltrials.gov/large-docs/19/NCT04012619/Prot_SAP_000.pdf